CLINICAL TRIAL: NCT00747019
Title: Prosocial Behavior and Exercise Among Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Capri G. Foy, Ph.D., M.S, Division of Public Health Sciences, Wake Forest University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: AG0106; 1R21AG027413-01A2 (NIH)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Health-Related Quality of Life; Physical Activity; Physical Function
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PBPA (Experimental)
  Interventions: Behavioral: Prosocial Behavior Physical Activity (PBPA)
- PE (Active Comparator)
  Interventions: Behavioral: Physical Exercise (PE)

INTERVENTIONS:
Behavioral: Prosocial Behavior Physical Activity (PBPA) — The PBPA condition involves a center-based cognitive-behavioral intervention to teach participants the behavioral skills to engage in long-term (9-month) independent physical activity; delivered three times a week months 1-3; independent physical activity months 4-9. PBPA participants also earn boxes of food for donation to the Second Harvest Food Bank (SHFB) of Northwest North Carolina based upon their weekly physical activity.
  Arms: PBPA
Behavioral: Physical Exercise (PE) — The PE condition is a center-based cognitive-behavioral intervention to teach participants the behavioral skills to engage in long-term (9-month) independent physical activity; delivered three times a week months 1-3; independent physical activity months 4-9.
  Arms: PE

SUMMARY:
The purpose of this study is to compare two exercise programs to determine how well they help older adults make exercise a regular habit after 9 months.

DETAILED DESCRIPTION:
Although only a small percentage of older adults engage in habitual physical activity, previous studies have demonstrated interventions that include cognitive-behavioral strategies can enhance long-term, independent physical activity. In addition, there are episodic charity events, such as charity walks, that attract large numbers of participants of all age ranges to engage in moderate-intensity physical activity. These actions are a form of prosocial behavior, defined as voluntary, intentional behavior that results in benefits for another. The opportunity to help others seems to be a motive in inspiring these individuals to at least engage in one session of moderate physical activity. Thus, the current research project contemplates whether prosocial behavior may be implemented as a viable behavioral incentive for long-term physical activity.

Both the Prosocial Behavior Physical Activity (PBPA) group and the Physical Exercise (PE) group will receive a cognitive-behavioral intervention to teach participants the behavioral skills necessary to engage in long-term (9-month) independent physical activity. Both programs will provide supervised exercise sessions so that participants learn how to safely and effectively engage in physical activity, and both programs will help participants set goals for activity and overcome barriers to exercise. However, in PBPA group, participants will be able to also earn boxes of food for donation to a charity based upon their physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Between 55 and 80 years of age
* Physically underactive (moderate or vigorous physical activity for less than 2 days per week for the preceding 3 months)
* No evidence of any major psychological illness
* Written permission from the participant's primary care physician with specific certification of no severe risk of cardiovascular disease
* Participant resides within a 35-mile radius of the study site
* Participant will remain in the area for the duration of the study

Exclusion Criteria:

* Self-reported evidence of cardiovascular disease risk, or documentation by the primary care physician of at least one of the following within the past 5 years:

  * Myocardial infarction (MI)
  * Percutaneous transluminal coronary angioplasty (PTCA)
  * Chronic or unstable angina at rest or during physical exertion
  * New York Heart Association (NYHA) Type I through Type IV congestive heart failure
  * Unstable ventricular arrhythmias
  * Cardiovascular surgery (coronary artery or valvular heart disease)
  * Ischemic or hemorrhagic stroke
  * Intermittent claudication during physical activity
  * Edema in feet
* Self-reported or documented evidence of rheumatoid arthritis
* Self-reported or physician-reported evidence of current cigarette or cigar smoking
* Self-reported treatment for psychiatric illness within the past 5 years:

  * Treatment for major depression or schizophrenia
  * Currently receiving lithium or neuroleptics
  * Hospitalization with the last 5 years for depression, or clinical judgment of treatment for major depression
* Hearing or sight impairments
* Cognitive impairment
* Alcohol consumption greater than 21 drinks per week, or self-reported alcoholism
* Inability to speak or read English
* Judgment of clinical staff
* Current participation in another medical intervention study

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Self-reported physical activity | Baseline, 3 and 9 months

SECONDARY OUTCOMES:
Physical function, health-related quality of life | Baseline, 3 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Capri G. Foy, PhD, MS, Principal Investigator — Division of Public Health Sciences, Wake Forest University School of Medicine
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Rejeski WJ, Brawley LR, Ambrosius WT, Brubaker PH, Focht BC, Foy CG, Fox LD. Older adults with chronic disease: benefits of group-mediated counseling in the promotion of physically active lifestyles. Health Psychol. 2003 Jul;22(4):414-23. doi: 10.1037/0278-6133.22.4.414. PMID 12940398
- [Background] Rejeski WJ, Foy CG, Brawley LR, Brubaker PH, Focht BC, Norris JL 3rd, Smith ML. Older adults in cardiac rehabilitation: a new strategy for enhancing physical function. Med Sci Sports Exerc. 2002 Nov;34(11):1705-13. doi: 10.1097/00005768-200211000-00003. PMID 12439072
- [Background] Eisenberg N, Miller PA. The relation of empathy to prosocial and related behaviors. Psychol Bull. 1987 Jan;101(1):91-119. No abstract available. PMID 3562705